CLINICAL TRIAL: NCT01791569
Title: Sensor Off Studies Using a Bedside Respiratory Patient Monitoring System With the Multi-Functional Patient Monitoring PCBA-1
Brief Title: Pulse Oximetry- Evaluating Sensor Off- PCBA-1
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPR0303
Record Dates: First submitted 2012-11-29; First posted 2013-02-15 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2013-12

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To demonstrate that the sensor-off feature on the Pulse oximeter displays per specifications when the sensor is removed from the finger.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 or older (inclusive).
2. Subject is able to participate for the duration of the study
3. Subject is willing to sign an informed consent

Exclusion Criteria:

1. Previous injury or trauma to fingers or hands that may change blood flow or vascular supply and affect our ability to test sensors
2. Physiologic abnormalities that prevent proper application of a medical sensor and electrode
3. Severe contact allergies that cause a reaction to standard adhesive materials such as those found in medical sensors and electrodes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy, Well Perfused subjects
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Device posts Sensor Off within 1 minute after sensor is removed at least 90% of the time. | 1-2 hours per subject

CONTACTS AND LOCATIONS:
Locations (1):
- Covidien, Boulder, Colorado, United States